CLINICAL TRIAL: NCT00841204
Title: Phase II Trial of Sulindac in Individuals at Increased Risk for Melanoma
Brief Title: Sulindac in Preventing Melanoma in Healthy Participants Who Are at Increased Risk of Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-01115; NCI-2009-01115 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UARIZ-08-0841-04; CDR0000633938; N01CN35158 (NIH); 08-0841-04 (Other: University of Arizona Health Sciences Center); UAZ05-2-10 (Other: DCP); P30CA023074 (NIH)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Precancerous Condition
MeSH Terms: conditions — Precancerous Conditions | interventions — Sulindac

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Experimental): Participants receive oral sulindac twice daily for 8 weeks
  Interventions: Drug: sulindac; Other: laboratory biomarker analysis
- Arm II (Placebo Comparator): Participants receive oral placebo twice daily for 8 weeks
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sulindac — Given orally
  Other Names: Aflodac; Algocetil; Clinoril; SULIN
  Arms: Arm I
Other: placebo — Inactive agent
  Other Names: PLCB
  Arms: Arm II
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well sulindac works in preventing melanoma in healthy participants who are at increased risk of melanoma. Sulindac may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether sulindac is more effective than a placebo in preventing melanoma in individuals with many moles and abnormal moles.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine sulindac and metabolite levels in healthy participants with atypical nevi and benign nevus at increased risk for melanoma treated with sulindac versus placebo.

SECONDARY OBJECTIVES:

I. To assess the effects of sulindac on apoptosis in atypical nevi of these participants.

II. To assess the effects of sulindac on VEGF expression in atypical nevi of these participants.

III. To assess sulindac and metabolite levels in plasma and its association with drug levels in the target tissue.

OUTLINE: This is a multicenter study. Participants are randomized to 1 of 2 treatment arms.

ARM I: Participants receive oral sulindac twice daily.

ARM II: Participants receive oral placebo twice daily.

In both arms, treatment continues for 8 weeks in the absence of unacceptable toxicity.

Blood and tissue samples are collected at baseline and/or after completion of study therapy and analyzed for sulindac and metabolite levels via high performance liquid chromatography tandem mass spectrometry; the detection of apoptotic cells via TUNEL assay; and VEGF expression via immunohistochemistry assays.

After completion of study therapy, participants are followed for 2 weeks.

ELIGIBILITY:
Criteria:

* Healthy participants at risk for developing melanoma and meeting the following criteria: must have >= 4 large (>= 5 mm and < 15 mm) atypical nevi and have 1 benign nevus amenable to biopsies
* No histologically confirmed melanoma on the baseline biopsy
* No more than 1 prior cutaneous melanoma
* One prior stage I, IIA, or IIB melanoma allowed provided patients have been off treatment > 3 months
* Modified dermoscopy score < 4.8
* Karnofsky performance status 80-100%
* ANC >= 1,500/mm^3
* No family history of melanoma involving >= 2 first degree relatives
* Platelets count >= 100,000/mm^3
* Total bilirubin =< 2.0 mg/dL
* AST/ALT =< 2.0 times upper limit of normal
* Creatinine =< 1.5 mg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception
* More than 6 months since prior and no concurrent tanning bed use or other methods to promote sun-tanning
* Willing to minimize sunlight exposure by applying sunscreen/sunblock or wearing clothing to shield skin during outdoor activity during study participation
* Willing or able to limit alcohol consumption to less than 3 servings a week during the study period
* No frequent, chronic or moderate/severe gastrointestinal (GI) complaints
* Upper GI problems requiring prescription or nonprescription medical remedies for symptoms of heartburn, dyspepsia, nausea, or abdominal pain > once a week on average
* History of peptic ulcer, occult or gross intestinal bleeding
* No prior allergic reaction to aspirin (unless subsequent dosing with other NSAIDs has been well tolerated)
* No history of allergic reaction to lidocaine or xylocaine
* No history of allergic reaction (e.g., urticaria, asthma, or rhinitis) or gastric intolerance attributed to compounds of similar chemical or biological composition to sulindac
* No invasive cancer or cancer treatment within the past 5 years, except nonmelanoma skin cancer
* No immunosuppression by medication or disease, including any of the following: AIDS, oral prednisone, immunosuppressant/immunomodulator (i.e., cyclosporine, chemotherapeutic agent, or biologic therapy)
* No uncontrolled intercurrent illness
* No ongoing or active infection
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No psychiatric illness/social situations that would limit compliance with study requirements
* At least 30 days since prior participation and no concurrent enrollment or planning to enroll in another clinical trial
* No NSAIDs for more than 5 days per month within the past 3 months and no concurrent non-study NSAIDs, except low dose aspirin (81 mg/day)
* Willing or able to refrain from herbal medicines, above-standard vitamins, or minerals during study
* Standard daily multivitamin/mineral supplement (i.e., therapeutic doses of calcium and vitamin D for osteoporosis) allowed
* No concurrent lithium, phenytoin, or sulfonamides
* WBC >= 3,000/mm^3
* No history of bleeding or clotting disorder
* At least 3 months since prior and no concurrent coumadin or other systemic anticoagulant other than aspirin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Hui (Sherry) Chow, Principal Investigator — University of Arizona Health Sciences Center
Locations (2):
- United States (2):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Stanford University Hospitals and Clinics, Stanford, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Sulindac: Participants receive oral sulindac twice daily for 8 weeks in the absence of unacceptable toxicity.
- Placebo: Participants receive oral placebo twice daily for 8 weeks in the absence of unacceptable toxicity.
Period: Overall Study
Arm/Group | Sulindac | Placebo
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulindac | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.0) | 45.9 (8.59) | 46.0 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 13 | 15 | 28
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Sulindac Concentration in the Nevi (Moles)
Time Frame: 8 weeks
Population: All randomized participants were included in the analysis except one participant in the sulindac arm did not provide nevi sample for analysis
Measure: Mean (Standard Deviation); unit: µg/g tissue
Arm/Group | Sulindac | Placebo
Number analyzed (Participants) | 24 | 25
µg/g tissue | 0.51 (1.05) | 0 (0)

2. Primary Outcome: Sulindac Sulfone, an Active Metabolite of Sulindac, Concentration in the Nevi
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/g tissue
Arm/Group | Sulindac | Placebo
Number analyzed (Participants) | 24 | 25
µg/g tissue | 1.38 (2.86) | 0 (0)

3. Primary Outcome: Sulindac Sulfide, an Active Metabolite of Sulindac, Concentration in the Nevi
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/g tissue
Arm/Group | Sulindac | Placebo
Number analyzed (Participants) | 24 | 25
µg/g tissue | 0.12 (0.12) | 0 (0)

4. Secondary Outcome: Sulindac Effects on Apoptosis in Atypical Nevi
Description: Change in the expression of a marker of apoptosis, cleaved caspase 3, in melanocytic junctional component
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: % of stained cells * intensity score
Arm/Group | Sulindac | Placebo
Number analyzed (Participants) | 20 | 21
% of stained cells * intensity score | 3 [-8 to 32] | -25 [-55 to -10]
Statistical Analysis 1: Comparison: Sulindac vs Placebo; Test type: Other; p = 0.0056, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Sulindac Effects on Vascular Endothelial Growth Factor (VEGF) Expression in Atypical Nevi
Description: Change in VEGF expression in melanocytic junctional component
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: % of stained cells * intensity score
Arm/Group | Sulindac | Placebo
Number analyzed (Participants) | 20 | 21
% of stained cells * intensity score | 23 [-13 to 50] | 0 [-50 to 35]
Statistical Analysis 1: Comparison: Sulindac vs Placebo; Test type: Other; p = 0.386, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Association Between Plasma and Target Tissue Sulindac Levels
Time Frame: 8 weeks
Population: The correlation between plasma and target tissue sulindac levels was analyzed for Arm I only because participants in Arm 2 did not have any measurable drug levels.
Measure: Number; unit: correlation coefficient
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 24 | 0
correlation coefficient | 0.41 |
Statistical Analysis 1: Comparison: Arm I; Test type: Other; p < 0.05, Regression, Linear

7. Secondary Outcome: Association Between Plasma and Target Tissue Sulindac Sulfone Levels
Time Frame: 8 weeks
Population: The correlation between plasma and target tissue sulindac sulfone levels was analyzed for Arm I only because participants in Arm 2 did not have any measurable drug levels.
Measure: Number; unit: correlation coefficient
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 24 | 0
correlation coefficient | 0.13 |
Statistical Analysis 1: Comparison: Arm I; Test type: Other; p = 0.58, Regression, Linear

8. Secondary Outcome: Association Between Plasma and Target Tissue Sulindac Sulfide Levels
Time Frame: 8 weeks
Population: The correlation between plasma and target tissue sulindac sulfide levels was analyzed for Arm I only because participants in Arm 2 did not have any measurable drug levels.
Measure: Number; unit: correlation coefficient
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 24 | 0
correlation coefficient | 0.33 |
Statistical Analysis 1: Comparison: Arm I; Test type: Other; p = 0.12, Regression, Linear

ADVERSE EVENTS:
Arm/Group | Sulindac | Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 22/25 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulindac (N=25) | Placebo (N=25)
Vasovagal episode (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sulindac (N=25) | Placebo (N=25)
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0
Heartburn (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 5 | 1
Prutitus (Skin and subcutaneous tissue disorders) | 2 | 3
Other skin disorders (Skin and subcutaneous tissue disorders) | 2 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 2
Allergic reaction (Immune system disorders) | 1 | 2
Sinus infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Other infection (Infections and infestations) | 4 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Extremity/Limb pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Nasal/Paranasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Larynx/Pharynx/Throat pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 0 | 2
Uterus pain (Reproductive system and breast disorders) | 4 | 2
Skin pain (Skin and subcutaneous tissue disorders) | 4 | 3
Fatigue (General disorders) | 3 | 3
Fever (General disorders) | 2 | 0
Headache (Nervous system disorders) | 14 | 14
Flu-like syndromes (General disorders) | 5 | 5
Other pain (General disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less